CLINICAL TRIAL: NCT03344510
Title: Kinetic Anesthesia Device for Lidocaine Injection: a Randomized Split-body Study of the Effects of Kinetic Anesthesia Devices on Pain of Lidocaine Injection in Healthy Volunteers
Brief Title: Kinetic Anesthesia Device Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Joseph F Sobanko M.D., Assistant Professor, Dermatology, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 828686
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Local Anaesthetic Complication; Pain
Keywords: lidocaine; vibration; anesthesia; injection; pain; discomfort; dermatology; dermatologic surgery; local; device
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study will be an open label split-body crossover trial, using healthy adult volunteers recruited from the faculty, staff and student body of the University of Pennsylvania, and from the University City area of Philadelphia. Participants will be randomized to one of three anatomic sites deemed relevant: the nasofacial sulcus, the lateral forehead, and the upper back. Participants will then be randomized to receive injection with the KAD first or second. They will receive one injection with and one injection without the interventional device, in a randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Kinetic anesthesia device, then no intervention (Experimental): In this arm of the crossover study, participants will receive lidocaine injection in conjunction with the kinetic anesthesia device, then will receive an injection without the kinetic anesthesia device intervention
  Interventions: Device: Kinetic Anesthesia Device; Other: Control
- No intervention, then kinetic anesthesia device (Experimental): In this arm of the crossover study, participants will receive lidocaine injection without the kinetic anesthesia device intervention, then will receive an injection in conjunction with the kinetic anesthesia device.
  Interventions: Device: Kinetic Anesthesia Device; Other: Control

INTERVENTIONS:
Device: Kinetic Anesthesia Device — A vibrating device held to the skin in close proximity to the lidocaine injection, intended to diminish discomfort by the gate control theory of pain
Other: Control — One injection will be administered without the kinetic anesthesia device.

SUMMARY:
Patients experience discomfort from lidocaine injections. Vibrating kinetic anesthesia devices (KAD) have been shown to reduce pain of injections in dentistry, pediatrics, and dermatology, though no studies of lidocaine injections in sites common to dermatologic surgery exist. We will conduct a randomized split-body study, in which healthy volunteers will rate the pain of lidocaine injections on a visual analog scale, with and without the vibrating kinetic anesthesia device being used during injection

DETAILED DESCRIPTION:
The study will be an open label split-body crossover trial, using healthy adult volunteers recruited from the faculty, staff and student body of the University of Pennsylvania, and from the University City area of Philadelphia. Participants will be randomized to one of three anatomic sites deemed relevant: the nasofacial sulcus, the lateral forehead, and the upper back. Participants will then be randomized to receive injection with the KAD first or second. The injection will be 0.5 cc of room temperature buffered lidocaine injected at constant slow speed (approximately 5 seconds) through a 30-gage needle held perpendicular to the skin by the same surgeon, with verbal cues standardized. Injections will be given in accordance with the standard of practice. When the KAD is used it will be used as directed: firmly pressed on the skin adjacent to the injection, with the needle aimed into the lighted area. Volunteers will evaluate each injection immediately after it is complete using the visual analog scale. When both injections are completed, participants will indicate their preference of injection, complete qualitative questions, and note necessary demographic information. Injection location and order of intervention (i.e. first or second) will be noted.

ELIGIBILITY:
Inclusion Criteria:

1. Adult volunteers greater than or equal to 18 years of age
2. Able and willing to provide informed consent
3. Able to comprehend and comply with study instructions, and able to complete necessary evaluations.

Exclusion Criteria:

1. Patients unable or unwilling to provide informed consent.
2. Patients with lidocaine allergy
3. Patients with known pain-related or neurological condition.
4. Patients with a known cardiac condition
5. Vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-01-27 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Sobanko, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were recruited from the area surrounding the University of Pennsylvania using IRB-approved flyers, as well as approved email communications, and postings on an approved website
Pre-assignment Details: This was a split body study, so each participant functioned in both intervention and control arms.
Period: First Injection (5 Minutes)
Arm/Group | Kinetic Anesthesia Device, Then no Intervention | No Intervention, Then Kinetic Anesthesia Device
Started | 21 | 26
Received Injection | 21 | 26
Completed | 21 | 26
Not Completed | 0 | 0
Period: Wash Out (10 Minutes
Arm/Group | Kinetic Anesthesia Device, Then no Intervention | No Intervention, Then Kinetic Anesthesia Device
Started | 21 | 26
Completed | 21 | 26
Not Completed | 0 | 0
Period: Second Injection (5 Minutes)
Arm/Group | Kinetic Anesthesia Device, Then no Intervention | No Intervention, Then Kinetic Anesthesia Device
Started | 21 | 26
Received Injection | 21 | 26
Completed | 21 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was a split body study, meaning that each participant was a part of both the "KAD" arm and the control arm.
Groups:
- All Participants: All participants received two lidocaine injections - one on the left and one on the right side of the body, with the left side injection always administered first. One of the injections was performed with the kinetic anesthesia device assistance, while the other was performed without (the control injection).
  As noted in the protocol, participants were randomized to receive the kinetic anesthesia device assisted injection first or second. 21 participants received the kinetic anesthesia device assisted injection first, while 26 were randomized to receive it second.
  Kinetic Anesthesia Device: A vibrating device held to the skin in close proximity to the lidocaine injection, intended to diminish discomfort by the gate control theory of pain
Arm/Group | All Participants
Number analyzed (Participants) | 47
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [23 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Self-identified race and ethnicity: White (non-hispanic) | 20
  Self-identified race and ethnicity: Asian | 13
  Self-identified race and ethnicity: White (hispanic) | 8
  Self-identified race and ethnicity: African-American | 5
  Self-identified race and ethnicity: Native American | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain of Lidocaine Injection, Measured by Visual Analog Scale.
Description: Participants will be asked to mark the pain of injection on a 100mm visual analog scale. The visual analog scale is commonly used to measure acute pain, though it can be used in other settings. It consists of a line 100mm long. The left end is labeled "no pain at all" and the right end is labeled "worst pain imaginable." Participants will rate pain by marking the scale where they feel that their level of pain falls on the scale. The length from 0 to the participant's mark will be measured in millimeters (for a range of 0 to 100 mm possible). Higher numbers will be considered more pain.
Time Frame: This measurement will occur immediately after each injection
Population: See above
Measure: Median (Inter-Quartile Range); unit: mm on visual analog scale
Groups:
- Injections Using the Kinetic Anesthesia Device: Participants graded the pain of lidocaine injection perfomed in conjunction with the kinetic anesthesia device
  Kinetic Anesthesia Device: A vibrating device held to the skin in close proximity to the lidocaine injection, intended to diminish discomfort by the gate control theory of pain
- Injections Without Kinetic Anesthesia Device: Participants graded the pain of lidocaine injection with no intervention
Arm/Group | Injections Using the Kinetic Anesthesia Device | Injections Without Kinetic Anesthesia Device
Number analyzed (Participants) | 47 | 47
mm on visual analog scale | 7.5 [5 to 16] | 26 [13 to 34]

2. Secondary Outcome: Patient Preference for Injection With or Without Kinetic Anesthesia Device
Description: Qualitative measure of patient preference for injections with or without the kinetic anesthesia device.
  Participants were asked whether they preferred the injection with or without the kinetic anesthesia device.
  Counts below indicate the number of participants who preferred each type of injection.
Time Frame: This will occur immediately after the second injection
Population: 45 participants filled out this portion of the post-injection questionnaire, while two neglected this portion of the questionnaire.
Measure: Count of Participants; unit: Participants
Groups:
- Kinetic Anesthesia Device Injection: Participants received the lidocaine injection in conjunction with the kinetic anesthesia device
  Kinetic Anesthesia Device: A vibrating device held to the skin in close proximity to the lidocaine injection, intended to diminish discomfort by the gate control theory of pain
- Control Injection: Participants received lidocaine injection with no intervention
Arm/Group | Kinetic Anesthesia Device Injection | Control Injection
Number analyzed (Participants) | 45 | 45
Participants | 33 | 6

ADVERSE EVENTS:
Time Frame: 1 Hour
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT03344510/Prot_SAP_000.pdf